CLINICAL TRIAL: NCT04874961
Title: Olive Polyphenols in Cardiovascular Prevention: Efficacy and Tolerability of a Commercially Available Standardized Olive Extract (Tensiofytol®) as Compared to Placebo in Patients With Elevated Blood Pressure: a RDBPC Trial.
Brief Title: Olive Polyphenols in Cardiovascular Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nina Hermans (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Sponsor-Investigator, Nina Hermans, Professor, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Olijfstudie 2021
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-01

CONDITIONS: Hypertension, Systolic
MeSH Terms: conditions — Isolated Systolic Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized olive extract (Tensiofytol®) (Experimental): 3 capsules/day during dinner Per day: 334 mg olive leave dry extract and 106 mg olive fruit dry extract (Olea europaea L.), equivalent to 100 mg oleuropein and 20 mg hydroxytyrosol
  Interventions: Dietary Supplement: Tensiofytol®
- Placebo (Placebo Comparator): 3 capsules/day during dinner
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Tensiofytol® — standardized olive extract
  Arms: Standardized olive extract (Tensiofytol®)
Other: Placebo — contains excipients only
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate whether the use of a commercially available standardized olive extract (Tensiofytol®) in individuals with elevated blood pressure

1. Leads to a clinically relevant reduction of blood pressure on the short term,
2. Leads to a clinically relevant reduction of cholesterol levels, especially LDL,
3. Leads to a change in oxidative stress biomarkers.

Participants will be stratified by sex before randomization to one of the three treatments for 8 weeks:

* Tensiofytol: 100 mg oleuropein and 20 mg hydroxytyrosol per day
* Placebo

All treatments have an identical shape and color and should be used in the same way (oral intake; 3 capsules/day during dinner). No dietary instructions are given and participants are asked not to change their dietary habits, nor to start other therapies (medication, supplements, slimming diets, extra physical activity, etc.) during their study period. Standardized questionnaires are used to obtain information on demographics, dietary habits and side effects. At baseline and after 8 weeks, 27 ml blood is drawn for various biological analyses, and blood pressure, BMI and waist circumference are measured.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure ≥ 130 mmHg

Exclusion Criteria:

* <18 jaar
* >76 jaar
* Smoking
* Use of nutritional supplements or (chronic) medication*
* Triglycerides > 400 mg/dL
* > 14 alcoholic consumptions/week
* Chronic illness (e.g. diabetes, atherosclerosis, reumatoid arthritis)
* Acute infection
* Current pregnancy or pregnancy wish during the study period
* Breast feeding

  * When nutritional supplements were used regularly, participation is allowed after a 10-day wash out period.

Use of medication will be individually assessed and is permitted if it does not interfere with the used treatments and the patient is stable on the medication.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline Blood Pressure, Systolic at 8 weeks | Baseline, 8 weeks
  average of 3 measurements during 15 minutes

SECONDARY OUTCOMES:
Frequency of side effects (+ their burden) as reported in the final questionnaire | 8 weeks
  Unvalidated but standardized questionnaire on typical statin-related side effects
Change from baseline Blood Pressure, diastolic at 8 weeks | Baseline, 8 weeks
  average of 3 measurements during 15 minutes
Change from baseline Blood Pressure, systolic at 4 weeks | Baseline, 4 weeks
  average of 3 measurements during 15 minutes
Change from baseline LDL cholesterol level at 8 weeks | Baseline, 8 weeks
  Calculated from Total Cholesterol, HDL Cholesterol and Triglycerides
Change from baseline HDL cholesterol level at 8 weeks | Baseline, 8 weeks
  Measurement in Serum
Change from baseline non-HDL cholesterol level at 8 weeks | Baseline, 8 weeks
  Calculated from HDL and total cholesterol
Change from baseline total cholesterol level at 8 weeks | Baseline, 8 weeks
  Measurement in Serum
Change from baseline triglycerides level at 8 weeks | Baseline, 8 weeks
  Measurement in Serum
Change from baseline Apo A1 level at 8 weeks | Baseline, 8 weeks
  Measurement in Serum
Change from baseline Apo B level at 8 weeks | Baseline, 8 weeks
  Measurement in Serum
Change from baseline lipoprotein A (LP(a)) level at 8 weeks | Baseline, 8 weeks
  Measurement in Serum
Change from baseline OxLDL level at 8 weeks | Baseline, 8 weeks
  Measurement with ELISA
Change from baseline gluathion (GSH) level at 8 weeks | Baseline, 8 weeks
  Measurement with in house HPLC method
Change from baseline malondialdehyde (MDA) level at 8 weeks | Baseline, 8 weeks
  Measurement with ELISA
Change from baseline Remnant Cholesterol at 8 weeks | Baseline, 8 weeks
  Calculated from total, HDL and LDL cholesterol

OTHER OUTCOMES:
Change from baseline insuline level at 8 weeks | Baseline, 8 weeks
  Required to correctly interpret glucose levels, Measurement in Serum
Change from baseline homocysteine level at 8 weeks | Baseline, 8 weeks
  Measurement in Homocysteine Serum
Change from baseline hs-CRP level at 8 weeks | Baseline, 8 weeks
  Measurement in Serum
Change from baseline creatinine level at 8 weeks | Baseline, 8 weeks
  Required to correctly interpret HbAc1 levels, Measurement in Serum
Change from baseline HbA1c level at 8 weeks | Baseline, 8 weeks
  Measurement in EDTA Whole Blood
Change from baseline hemoglobine level at 8 weeks | Baseline, 8 weeks
  Required to correctly interpret HbAc1 levels, Measurement in EDTA Whole Blood
Change from baseline creatine kinase (CK) level at 8 weeks | Baseline, 8 weeks
  Measurement in serum
Change from baseline C-peptide level at 8 weeks | Baseline, 8 weeks
  Measurement in serum
Change from baseline waist circumference at 8 weeks | Baseline, 8 weeks
  Measurement with measuring tape
Change from baseline Body Mass Index (BMI) at 8 weeks | Baseline, 8 weeks
  weight and height will be combined to report BMI in kg/m^2
Change from baseline glucose level at 8 weeks | Baseline, 8 weeks
  Measurement in Fluoride Plasma

CONTACTS AND LOCATIONS:
Overall Officials: Johan Bosmans, Prof. MD., Principal Investigator — University Hospital, Antwerp
Locations (1):
- UAntwerp, NatuRAPT, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: No